CLINICAL TRIAL: NCT02245607
Title: Compensatory Cognitive Training in Clinical High Risk Latino Youth
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of California, San Diego (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Kristin Cadenhead, M.D., Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MH105247; 5R34MH105247-03 (NIH)
Record Dates: First submitted 2014-09-16; First posted 2014-09-19 (Estimated); Last update posted 2021-02-08 (Actual); Status verified 2021-02

CONDITIONS: Clinical High Risk; Psychosis; Prodromal; Schizophrenia
Keywords: Psychotic Disorders; Cognitive Training; Mental Disorders; Schizophrenia and Disorders with Psychotic Features
MeSH Terms: conditions — Psychotic Disorders; Schizophrenia; Mental Disorders; Schizophrenia Spectrum and Other Psychotic Disorders | interventions — Recreation Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Compensatory Cognitive Training (Experimental): Compensatory Cognitive Training
  Interventions: Behavioral: Compensatory Cognitive Training
- Recreational Therapy (Active Comparator): Recreational Therapy
  Interventions: Behavioral: Recreational Therapy

INTERVENTIONS:
Behavioral: Compensatory Cognitive Training
  Arms: Compensatory Cognitive Training
Behavioral: Recreational Therapy
  Arms: Recreational Therapy

SUMMARY:
This is a randomized study to compare Compensatory Cognitive Training (CCT) versus Recreational Therapy (RT) in Latino clinical high risk individuals in the US and Mexico.

Study hypotheses: Compared to those who receive RT, study participants receiving CCT will show significant improvement in neurocognition, functional capacity, self-rated functioning and clinical measures.

DETAILED DESCRIPTION:
This is a 12 week randomized study to compare Compensatory Cognitive Training (CCT) versus Recreational Therapy (RT) in Latino clinical high risk individuals in the US and Mexico.

Study participants will be measured 3 times, at baseline, 12 and 24 weeks on all outcome measures. Study hypothesis: Study participants receiving CCT will show significant improvement at 12 and 24 weeks compared to baseline in 1) Neurocognition using the Global Cognitive Index z score derived from the MATRICS neurocognitive domain scores, 2) Functional Capacity as assessed by the UCSD Performance-based Skills Assessment (UPSA/UPSA-Adolescent), 3) Self-Rated Functioning as measured by the Specific Level of Functioning Scale (SLoF) and 4) Clinical symptom ratings as measured by the Scale of Prodromal Symptoms (SOPS) total score when compared to subjects receiving RT training across study time.

ELIGIBILITY:
Inclusion Criteria:

* Meet Clinical High Risk criteria
* Be of Latino descent
* Speak Spanish as their preferred language

Exclusion Criteria:

* Concomitant medical or neurological illness
* Brain injury with loss of consciousness > 30 minutes
* Current substance abuse (excluding nicotine)
* IQ < 80
* High suicidal risk

Ages: 12 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2014-10; Primary Completion 2020-06-30 (Actual); Study Completion 2021-02-01 (Estimated)

PRIMARY OUTCOMES:
Neurocognition (Global Cognitive Index z score) | 3 and 6 months post-baseline
  The CGI is derived based on Z scores across multiple neurocognitive domains and is a representation of global cognition

SECONDARY OUTCOMES:
Functional capacity (UPSA/UPSA-A) | 3 and 6 month post-baseline
  The UPSA total Functional Capacity score is the total of all subscale scores on the UPSA (Finances, Communication, Transportation, Household)

OTHER OUTCOMES:
Self-reported functioning (SLoF) | 3 and 6 month post-baseline
  The specific level of functioning (SLOF) assessment scale measures observable behavioral functioning and daily living skills.
Clinical symptom severity (SOPS total) | 3 and 6 month post-baseline
  The Scale of Prodromal Symptoms (SOPS) measures positive, negative, disorganized and general symptoms seen in psychotic illness. The total score is used for outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Cadenhead, MD, Principal Investigator — University of California, San Diego
Locations (2):
- University of California San Diego, La Jolla, California, United States
- Instituto Nacional de Neurología y Neurocirugía, Mexico City, Mexico